CLINICAL TRIAL: NCT04439773
Title: Efficacy of Intravenous Infusion of Lidocaine in Sedation for ERCP: a Randomised Placebo-controlled Study
Brief Title: Intravenous Infusion of Lidocaine in Gastroscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2020SDU-QILU-022
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Sedation
Keywords: intravenous lidocaine gastroscopy bucking
MeSH Terms: interventions — Sodium Chloride; Lidocaine

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to controll group or lidocaine group. Participants of control group are given placebo while participants of lidocaine group are given lidocaine.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): the control group will be given the same volume of saline as the experimental group
  Interventions: Drug: placebo
- lidocaine group (Experimental): the experimental group will be given l-1.5mg lidocaine and then 2mg/kg/h
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: placebo — the control group will be given the same volume of saline.
  Other Names: saline
  Arms: control group
Drug: Lidocaine — the experimental group will be given 1-1.5mg/kg lidocaine and then 2mg/kg/h
  Other Names: Compound Lidocaine Hydrochloride Injiection
  Arms: lidocaine group

SUMMARY:
Intravenous infusion of lidocaine significantly reduces incidence of bucking when perfomed gastroscopy.

DETAILED DESCRIPTION:
This study divide patients into two groups, the patients in lidocaine group will be given lidocaine; the control group will be given placebo .the primary endopiont was to investigate whether intravenous lidocaine can reduce incidence of bucking and movement in sedation of gastroscopy.

ELIGIBILITY:
Inclusion Criteria:

patients aged >18 years who were scheduled for ERCP at Qilu hospital.

Exclusion Criteria:

patients with ASA (American Society of Anesthesiologists) Class 4 or 5, pre-existing hypoxemia (SpO2 <90%), hypotension (systolic blood pressure <90 mm Hg), bradycardia (HR<50 beats/min), uncontrolled hypertension (SBP >170 mm Hg, diastolic blood pressure>100 mm Hg), severe renal or liver failure, pregnancy or lactation, allergy to lidocaine, atrioventricular block, epilepsy, and inability to give informed consen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of bucking during the procedure | half a year
  the difference between incidence of bucking of the two groups

SECONDARY OUTCOMES:
propofol consumption difference between the two groups | half a year
  the total propofol dosage consumption between the two groups
the incidence of infusion pain when adminstrated propofol | half a year
  the infusion pain devied into no pain, mild pian, and severe pain
Safety assessed by the rate of hypoxia during the procedure | half a year
  Hypoxia, defined as peripheral oxygen saturation <90% for >30 seconds
Safety assessed by the rate of hypotention during the procedure | half a year
  Hypotension, defined as systolic blood pressure <90 mmHg
Safety assessed by the rate of breadycardia during the procedure | half a year
  Bradycardia, defined as heart rate <50 beats/min
Safety assessed by the rate of required airway management during the procedure | half a year
  Required airway management such as jaw lifting, mask ventilation, or tracheal intubation in severe hypoxia Required airway management such as jaw lifting, mask ventilation, or tracheal intubation in severe hypoxia
endoscopists satisfaction assessed by the performer | half a year
  the endoscopists satisfacition score were assessed on a 0-10VAS after the procedure
patient satisfaction assessed by the patient | half a year
  the patient satisfacition score were assessed on a 0-10VAS 30mins after the procedure
anesthetist satisfaction | half a year
  the anesthetist satisfacition score were assessed on a 0-10VAS 30mins after the procedure
pain socre after the gastroscopy | half a year
  pain were measured on a 0-10VAS at arrival in the recovery room ,30min later
fatigue score after the ERCP | half a year
  fatigue were measured on a 0-10VAS at arrival in the recovery room ,30min later

CONTACTS AND LOCATIONS:
Overall Officials: Shan dong China, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided